CLINICAL TRIAL: NCT02067741
Title: A Stratified, Multicenter Phase II Trial of Transdermal CR1447 (4-OH-testosterone) in Endocrine Responsive-HER2 Negative and Triple Negative-androgen Receptor Positive Metastatic or Locally Advanced Breast Cancer
Brief Title: CR1447 in Endocrine Responsive-HER2neg and TN-ARpos Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The SAKK board decided to prematurely end the life-long follow-up of the trial SAKK 21/12, as 90% of the patients have died.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 21/12; SNCTP000000389 (Other: SNCTP)
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Breast Adenocarcinoma; Breast Cancer
Keywords: Post-menopausal women; topical application CR1447; endocrine responsive-HER2neg breast cancer; triple negative-androgen receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 4,17 beta-dihydroxy-4-androstene-3-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum A - HER2neg BC RD - CR1447 (Experimental): Stratum A - patients with endocrine responsive-HER2neg BC
  Interventions: Drug: CR1447
- Stratum B - ARpos B - CR1447 (Experimental): Stratum B - patients with triple-negative and confirmed ARpos BC
  Interventions: Drug: CR1447

INTERVENTIONS:
Drug: CR1447 — 400 mg, corresponding to two 4 g stick packs applications twice daily
  Other Names: 4-OHT

SUMMARY:
SAKK 21/12 is a stratified, multicenter Phase II first in-human trial with transdermal CR1447 (4-OH-testosterone) and is directed to patients with endocrine responsive-HER2neg and TN-ARpos metastatic or locally advanced breast cancer.

The trial will be conducted in Switzerland with max. 90 patients. CR1447 has a very good safety and tolerability profile and combines two mechanisms of action, interaction with the AR and the aromatase enzyme may have a higher activity than drugs with a single mechanism and might offer the possibility of non-chemotherapy based endocrine therapy to the limited treatment options in TN-ARpos BC. Transdermal application of CR1447 might have the advantage to continuously release of 4-OHT into the blood stream, thus omitting a first pass effect.

In Phase II the main objective is to assess activity and to determine the efficacy and tolerability of CR1447. Phase II will consist of two strata, into which patients will be stratified according to their hormonal receptor status: Stratum A for patients with endocrine responsive-HER2neg disease, regardless of their AR status and Stratum B for patients with triple-negative and determined ARpos disease. Patients with triple-negative disease tested negative for AR will be excluded from the trial.

In both strata patients will be treated with 400 mg of CR1447 until disease progression, patients' wish or physicians' decision to end treatment. Biopsies of one defined metastatic lesion in those patients who gave informed consent will be performed at baseline and within the third week of treatment with CR1447.

Measurement of AR expression, expression of downstream targets of ERα, ERβ, PR, AR, angiogenesis and other translational studies as described in this protocol should help confirming the hypothesis of an increased benefit of CR1447 due to its dual action, efficacy of topical application, tolerability and in deciding whether one should proceed to a large randomized trial.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer and a heterogeneous disease and tumor categorization based on molecular characteristics beyond the currently used markers such as the estrogen receptor (ER), progesterone receptor (PR), and HER2, makes tumor categorization and treatment a demanding task.

The treatment and prevention of relapses of breast cancer is mainly based on I) surgery of primary tumors, II) radiotherapy, III) chemotherapy, IV) endocrine therapy, and V) specific interventions. Although there have been advances in breast cancer therapy with three out of four women with breast cancer now being cured, one out of four patients will relapse or present with metastatic disease at the time of first diagnosis and hence be incurable and die of their disease.

The endocrine responsive breast cancer is defined by the immunohistochemical detection of the ER (estrogen receptor) and/or the PR (progesterone receptor) on at least 1% of tumor cells on the tissue sample to a variable degree and offers the possibility of treatment using endocrine strategies in about 80% of patients. Endocrine responsive breast cancers may also express HER2. The triple negative breast cancer (TNBC) is defined by the lack of expression of ER, PR, and HER2. The analysis is made on the pathological tumor tissue sample. While for ER and PR, the threshold is less than 1% of tumor cells expressing both receptors, HER2 negativity is defined as immunohistochemical scores of 0/1+ or tumors with scores of 0/1+ or 2+ that are lacking HER2 gene amplification after in situ hybridization. Approximately 15% of all breast cancers are found to be triple-negative. However, due to the biologically more aggressive behavior of these tumors, the patient group suffering from this type of disease are overrepresented within the first five years after initial diagnosis.

Recently, androgen receptor (AR) targeted therapies gained new interest due to the fact that the AR is the most abundantly expressed sex hormone receptor in breast cancer (approx. 70% of all breast tumors) and, importantly, in about 20% (range 10% to 50% depending on the respective reference) of triple-negative breast tumors. The threshold for ARpos breast cancer is that >0% of tumor cells expresses the AR. In addition, a significant association was found between AR expression and longer overall survival of breast cancer patients. Androgens can induce proliferative changes in breast cancer cell lines, and testosterone acts as a tumor promoter in several animal models of breast cancer.

Endocrine responsive breast cancer Anti-estrogen therapy includes ovariectomy, to remove the primary source of female sex hormone in premenopausal women, and the application of luteinizing hormone releasing hormone (LHRH) agonists, to decrease the release of LH and prevent gonadal estrogen synthesis. These therapies induce a postmenopausal status. The hormonal treatment of choice for premenopausal women with ER positive metastatic breast tumors is the use of ER antagonists such as tamoxifen. Tamoxifen and aromatase inhibitors, preventing the final conversion of androgens to estrogens, are the main endocrine treatment options for postmenopausal women with metastatic breast cancer. The persisting estrogen levels in postmenopausal women are mainly due to aromatase activity in extragonadal sources such as breast tissue, skeletal muscle and adipose tissue. Thus, both ER blockade by tamoxifen and inhibition of estrogen synthesis inhibit the growth signal for breast cancer cells expressing ER.

Aromatase, the key enzyme of estrogen production in women, is expressed in and around breast tumors, in ovaries, and in skeletal muscle and adipose tissue in postmenopausal women. Several aromatase inhibitors (AI) have been developed. The first generation aromatase inhibitors include testolactone and aminogluthetimide that were replaced by the more potent second generation inhibitors fadrazole and formestane (4-hydroxy-4-androstenedione, 4-OHA), and later on by the even more potent third generation inhibitors exemestane, letrozole and anastrozole. 4OHA and exemestane are steroidal AI and irreversibly block aromatase while the non-steroidal AI letrozole and anastrozole are reversible inhibitors. Importantly, there seems to exist no cross-resistance between the two aromatase inhibitor classes, and 4-OHA or exemestane may still show efficacy after relapse upon letrozole/anastrozole treatment.

In summary, there is a great demand for novel and improved therapeutic strategies, especially to overcome resistance to chemotherapy or presently available endocrine therapy in postmenopausal women.

While patients with ER and/or PR positive tumors can be treated with endocrine therapies and patients with HER2pos disease with treatments directed against HER2 such as trastuzumab, lapatinib, and trastuzumab/pertuzumab combination therapy, no endocrine or targeted anti-HER2 directed therapy exists for patients suffering from triple negative disease.

For these patients, only chemotherapy is a therapeutic option. Unfortunately, these tumors tend to be aggressive and quickly growing with a high relapse rate even after intensive adjuvant chemotherapy. Due to the absence of estrogen receptors, endocrine therapy based on anti-estrogen intervention strategies must fail.

There are currently no suitable treatment options for patients with metastatic triple-negative breast tumors whose disease has failed to respond to chemotherapy. Thus, there is a great demand for novel and improved therapeutic strategies in this patient group and in all patients with acquired resistance to combat breast cancer.

Testosterone was already used extensively between the 1930s and 1960s for breast cancer treatment, with anecdotal tumor responses (especially bone metastases) seen in up to 20% of treated women. Side effects such as hirsutism and aggressive behavior as signs of virilization in treated women and the evidence that testosterone may be easily be converted to estrogens in the body led to the discontinuation of its use.

CR1447 (4-hydroxytestosterone [4-OHT]) is a steroidal small molecule which has two distinct properties, acting as a steroidal aromatase inhibitor (AI) and binding to the AR with high affinity (IC50 4.4 nM). In vitro studies indicate that human breast cancer cell lines are inhibited by CR1447 in their growth if they express the androgen receptor, while knock out of the AR abolishes this effect. A significant proportion of 4-OHT is converted to 4-OHA (4-hydroxyandrostenedione, formestane). In vivo 4-OHT and 4-OHA, form a redox system. 4-OHA is the 17-beta-oxidized isoform of CR1447. 4-OHA had previously been approved as an aromatase inhibitor for the treatment of BC via intramuscular (i.m.) injection (Formestane, Lentaron®) injection, but was discontinued by Novartis due to the development of oral aromatase inhibitors. Unlike testosterone, both compounds, 4-OHA and 4-OHT, are not converted to estrogens in vivo. Due to a high first pass effect after oral dosing, 4-OHA had to be administered parentally e.g. as an intramuscular injection. While this regimen was clinically effective, local side effects were a dose limiting issue.

A clinical feasibility study of transdermally applied 4-OHA showed that significant amounts of 4-OHA are absorbed by the skin. Intramuscular and transdermally (twice daily) applied 4-OHA achieved comparable the same plasma levels from day 3 on.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent before registration.
* Post-menopausal women
* Locally advanced or metastatic, histologically confirmed breast adenocarcinoma requiring therapy and not suitable for local treatment.

  * Stratum A: endocrine responsive-HER2neg BC, specifically: ERpos (≥1%), PRpos (≥1%), HER2neg; or ERpos(≥1%), PRneg, HER2neg
  * Stratum B: triple negative BC (ERneg (<1%), PRneg (<1%), HER2neg) and ARpos (>0%).
* Positive AR of the most recent formalin-fixed paraffin-embedded (FFPE) biopsy determined by central pathology (Stratum B only). Note: TNBC patients with only locally assessed ARpos (>0%) status are not allowed to enter the trial in Phase II.

  * Stratum A: Patients had 1 line of prior endocrine treatment for advanced disease with a treatment duration of ≥6 months and no evidence of progression at 6 months. No previous chemotherapy for advanced disease is allowed.
  * Stratum B: TN-ARpos BC patients had ≤2 lines of prior chemotherapy treatment for advanced disease.
* Patient is suitable for endocrine treatment.
* Presence of ≥1 measurable or evaluable lesion according to RECIST 1.1.
* Tumor assessment to be performed within 28 days before or on registration.
* Baseline PRO questionnaire (FACT-ES) has been completed (Phase II only).
* WHO performance status 0-1.
* Age ≥ 18 years.
* Adequate hematological values: hemoglobin ≥100 g/L, ANC ≥1.5x109/L, platelets ≥100x109/L.
* Adequate hepatic function: total bilirubin ≤1.5xULN, ALT ≤2.5xULN (except for liver metastases ≤5xULN).
* Adequate renal function: serum creatinine ≤1.5xULN.

Exclusion Criteria:

* Previous malignancy within 5 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Uncontrolled central nervous system (CNS) metastases, pulmonary carcinomatous lymphangiosis (i.e., >50% invasion), or liver metastases on >1/3 of the liver on ultrasound or computed tomography (CT).
* Unsuitable for endocrine therapy (e.g. due to rapidly progressing disease or impending 6.2.3complication).
* Indication for chemotherapy.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out PRO forms, or interfering with compliance for oral drug intake.
* Concurrent treatment with other experimental drugs in a clinical trial within 30 days prior to trial treatment start or other anti-cancer therapy within 14 days. Treatment with bisphosphonates/denosumab is allowed. Bisphosphonates/denosumab treatment had to be started at least 3 months before registration.
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes).
* Known hypersensitivity to trial drug(s) or hypersensitivity to any other component of the trial drugs.
* Local tumor relapse only that is amenable to surgical treatment.
* Previous treatment with formestane (4-OHA).
* Radiotherapy (RT) within 4 weeks prior to treatment start .
* Concurrent estrogen or progestin therapy in any formulation.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Disease control at 24 weeks (DC24) | at 24 weeks
  DC24 is obtained in a patient who achieves complete response (CR) or partial response (PR) within the first 24 ± 2 weeks of treatment or stable disease (SD) for at least 24 weeks after treatment start according to the RECIST 1.1 criteria.
  For patients without CR or PR and no PD before 24 weeks:
  * If the tumor assessment at 24 ± 2 weeks is missing but a later assessment shows SD, the patient will be counted as obtaining DC24.
  * If the tumor assessment at 24 ± 2 weeks is missing and there are no further tumor assessments or the subsequent assessment shows PD, the patient will be counted as not obtaining DC24.
  Tumor assessments showing CR or PR have to be confirmed after 4 weeks.

SECONDARY OUTCOMES:
Adverse events | 30 days after treatment discontinuation and thereafter monthly until all adverse events related to the trial drug have resolved
PK analysis of CR1447 | at baseline, 3 and 6 months of treatment
Estradiol levels during treatment | at baseline, 3 and 6 months of treatment
mRNA expression signature of downstream target genes of the ERα, ERβ, PR, AR and angiogenesis in biopsies | measured at baseline (day 0) and at treatment and within the third week of treatment
Ki67 expression | measured at baseline (day 0) and at treatment and within the third week of treatment
Disease control at 12 weeks (DC12) | at 12 ± 1 weeks
Change in tumor size at 12 weeks | at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Vetter, MD, Study Chair — Universitätsspital Basel; Beat Thürlimann, Prof, Study Chair — Cantonal Hospital of St. Gallen
Locations (13):
- Switzerland (13):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Oncocare / Klinik Engeried, Bern
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Frauenfeld / Brustzentrum Thurgau, Frauenfeld
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich

IPD SHARING:
Plan to Share IPD: No